CLINICAL TRIAL: NCT02550080
Title: A Phase IV, Randomised, Multicentre, Double-blind, Study to Evaluate the Clinical Utility of Prospective Genetic Screening (HLA-B*1301) for Susceptibility to Dapsone Hypersensitivity Syndrome
Brief Title: Clinical Utility Of Genetic Screening For HLA-B*1301, On Susceptibility To Dapsone Hypersensitivity Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Provincial Institute of Dermatology and Venereology (Other)
Collaborators: Shandong Provincial Hospital (Other Government); Jinan Central Hospital (Other); Shandong Qianfo Hospital (Unknown); Jinan Military General Hospital (Other); Qingdao Hiser Medical Group (Other); Liaocheng People's Hospital (Other); Dongying People's Hospital (Other); Jining First People's Hospital (Other); Dezhou People's Hospital (Other); Jinan City Dermatology Hospital Prevention and Treatment (Unknown); Linyi City Dermatology Hospital Prevention and Treatment (Unknown); Jining City Dermatology Hospital Prevention and Treatment (Unknown); Weifang City Dermatology Hospital Prevention and Treatment (Unknown); Laiwu City Dermatology Hospital Prevention and Treatment (Other); Rizhao City Dermatology Hospital Prevention and Treatment (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SDPIDV-DDS-001
Record Dates: First submitted 2015-08-20; First posted 2015-09-15 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Allergic Cutaneous Vasculitis; Urticaria; Psoriasis; Acne; Bullous Skin Diseases; Sterile Pustulosis; Leprosy; Pneumocystis Pneumonia
MeSH Terms: conditions — Vasculitis, Leukocytoclastic, Cutaneous; Urticaria; Psoriasis; Acne Vulgaris; Skin Diseases, Vesiculobullous; Leprosy; Pneumonia, Pneumocystis | interventions — Dapsone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The prospective genetic screening arm (Experimental): Prospective HLA-B*1301 screen before administrated treatment included dapsone
  Interventions: Drug: Dapsone; Genetic: HLA-B*1301
- The control arm (Active Comparator): No HLA-B*1301 screen before administrated treatment included dapsone
  Interventions: Drug: Dapsone

INTERVENTIONS:
Drug: Dapsone — For the HLA-B*1301 positive subjects, dapsone will not be administrated.
Genetic: HLA-B*1301 — The prospective genetic screening group will be tested before administrating dapsone
  Arms: The prospective genetic screening arm

SUMMARY:
This Study is to evaluate the utility of prospective HLA-B*1301 screening on the incidence of dapsone hypersensitivity syndrome (DHS) in 3130 previously Dapsone(DDS)-naive patients. Those patients include allergic cutaneous vasculitis, urticaria, psoriasis, acne, bullous skin diseases, sterile pustulosis, leprosy, pneumocystis pneumonia and any other patients who need dapsone administration. The study has two (co-primary) objectives: i) to determine if screening for HLA-B*1301 prior to DDS-containing treatment results in a lower incidence of clinically-suspected DHS versus current standard of care (no genetic screening) and ii) to determine if screening for HLA-B*1301 prior to DDS-containing treatment results in a significantly lower incidence of immunologically-confirmed DHS versus current standard of care (no genetic screening or patch testing). The study consists of up to a 5-day screening period, a randomised observation period (Day 1 through Week 6) and, for subjects experiencing a suspected DHS and a subset of DDS-tolerant subjects, an epicutaneous patch test (EPT) assessment period. Eligible subjects will be randomised to one of two study arms: a Current Standard of Care Arm (no prospective genetic screening: Control) and a Genetic Screening Arm (prospective genetic screening: Case). Subjects identified as HLA-B*1301 positive in the prospective Genetic Screening Arm will not receive dapsone and will be excluded from further study. Subjects who experience suspected DHS during the 6-week observation would be withdrawn from dapsone and undergo EPT patch testing 6 weeks later.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cutaneous vasculitis, urticaria, psoriasis, acne, bullous skin diseases, sterile pustulosis, leprosy, pneumocystis pneumonia and any other patients who need dapsone administration.
* Subjects are dapsone-naive.
* All subjects must have a clinical need for treatment with dapsone that precedes the decision to participate in the study.
* All subjects are willing to complete the 6-weeks period clinical trial.
* All subjects are written informed consent.

Exclusion Criteria:

* Has previously received Dapsone therapy.
* The subject or any of their healthcare providers is aware of the subjects HLA type.
* Has been diagnosed with Glucose-6-phosphate dehydrogenase deficiency or methemoglobin reductase deficiency
* Satisfies any contraindications or restrictions to Dapsone therapy as listed in the product labels.
* Current severe illness, including heart, liver and renal failure, major organ allograft, malignancy requiring parenteral chemotherapy that can not be discontinued for the duration of the trial, or any other conditions which, in the opinion of the Investigator, would make the patient unsuitable for the study.
* Any laboratory abnormality at Screening which, in the opinion of the Investigator, should preclude the subject's participation in the study [alanine aminotransferase (ALT), glutamic oxaloacetic transaminase(ALT), et al).
* Pregnant women or women who are breastfeeding.
* Subject is, in the opinion of the Investigator, unable to complete the 6 week Observation period and the EPT assessments as required.
* A positive result for HLA-B*1301 in those subjects randomised to the genetic screening arm.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3130 (Estimated)
Dates: Start 2015-07; Primary Completion 2018-12 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of clinically-suspected DHS during the 6-week observation period | 6 weeks
  The primary outcome measure will be the total number of clinically suspected Dapsone induced hypersensitivity syndrome during the 6-week observation period in both the prospective-screening group and control group, as reported by the DHS incidence (DHS patients/ total participants).
Incidence of immunologically-confirmed DHS during the 6-week observation period | 6 weeks
  The primary outcome measure will be the total number of immunologically confirmed Dapsone induced hypersensitivity syndrome during the 6-week observation period in both the prospective-screening group and control group, as reported by the DHS incidence (DHS patients/ total participants).

CONTACTS AND LOCATIONS:
Overall Officials: Furen Zhang, Study Chair — Shandong Provincial Institute of Dermatology and Venereology
Locations (1):
- Shandong Provincial Institute of Dermatology and Venereology, Jinan, Shandong, China